CLINICAL TRIAL: NCT04689776
Title: The Effectiveness of Dual Task Training in Elderly With Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201912EM016
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Cognitive Training; Exercise
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Frequency Dual-Task Training (HF) (Experimental): The participants of HF will receive a total of 36 training sessions, and each session will contain 90-120 minutes of training.
  Interventions: Behavioral: Dual-Task Training
- Low Frequency Dual-Task Training (LF) (Experimental): The participants of LF will receive a total of 12 training sessions, and each session will contain 90-120 minutes of training.
  Interventions: Behavioral: Dual-Task Training

INTERVENTIONS:
Behavioral: Dual-Task Training — The programs are based on dual-task trainings which contain cognitive training and exercise simultaneously. For physical exercise, we will design the programs that involve balance or strength training components in the aerobic exercises. In terms of cognitive training, we will design self-made teaching aids and board games to train different domains of cognitive functions. We plan to assess the participants before and after the intervention programs. We expect that elders receiving dual-task training will improve on outcome measures, and the group with more frequency will have better performance. The results of the study will provide evidence of interventions for elderly with cognitive decline, thereby reducing the burden on their caregivers and the cost of medical resource.

SUMMARY:
Cognitive decline is the impairment of memory, execution, or language. Early detection of the individuals who manifest cognitive decline and provide appropriate interventions may help reduce the burden of their caregivers and the medical expenses of the health-care system. Many studies have found that dual-task training combining cognitive training and exercise can improve cognitive function in older adults. However, it is yet not clear the appropriate frequency of the effective dual-task training for elderly with cognitive decline. Thus, this study aims to compare the intervention effects of high frequency sequential and low frequency dual-task training for elderly with cognitive decline.

DETAILED DESCRIPTION:
Cognitive decline is the impairment of memory, execution, or language. Early detection of the individuals who manifest cognitive decline and provide appropriate interventions may help reduce the burden of their caregivers and the medical expenses of the health-care system. Many studies have found that dual-task training combining cognitive training and exercise can improve cognitive function in older adults. However, it is yet not clear the appropriate frequency of the effective dual-task training for elderly with cognitive decline. Thus, this study aims to compare the intervention effects of high frequency sequential and low frequency dual-task training for elderly with cognitive decline.

We anticipate recruiting a total of 80 participants with cognitive decline. The participants will be assigned into 2 groups: high frequency dual-task training (HF) and low frequency dual-task training (LF) groups. The participants of HF will receive a total of 36 training sessions, and each session will contain 90-120 minutes of training. The participants of LF will receive a total of 12 training sessions, and each session will contain 90-120 minutes of training. The programs are based on dual-task trainings which contain cognitive training and exercise simultaneously. For physical exercise, we will design the programs that involve balance or strength training components in the aerobic exercises. In terms of cognitive training, we will design self-made teaching aids and board games to train different domains of cognitive functions. We plan to assess the participants before and after the intervention programs. We expect that elders receiving dual-task training will improve on outcome measures, and the group with more frequency will have better performance. The results of the study will provide evidence of interventions for elderly with cognitive decline, thereby reducing the burden on their caregivers and the cost of medical resource.

ELIGIBILITY:
Inclusion Criteria:

* able to follow instruction (MMSE>= 20)
* self- or informant-reported memory or cognitive complaint.

Exclusion Criteria:

* recent myocardial infarction,heart failure,recent heart surgery,
* severe asthma, concomitant with other neurological disorders, or joint deformity that might prevents them performing exercise or cognitive training.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change scores of the Montreal Cognitive Assessment (MoCA) | baseline, posttest (around 12 weeks after baseline)
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Change scores of Mini-Mental State Exam (MMSE) | baseline, posttest (around 12 weeks after baseline)
  The Mini-Mental State Examination (MMSE) is the most commonly administered psychometric screening assessment of cognitive functioning. The MMSE is used to screen patients for cognitive impairment, track changes in cognitive functioning over time, and often to assess the effects of therapeutic agents on cognitive function. The total score of MMSE ranged from 0 to 30. Higher values represent a better cognitive functioning.
Change scores of the Stroop test | baseline, posttest (around 12 weeks after baseline)
  The Stroop test will be used to assess the processing speed, inhibition, set-shifting, and selective attention abilities. The participants will be tested under 2 conditions: congruent and incongruent conditions. In the congruent condition, the color ink of a word is consistent with the written color name; while the color ink differs from the written color name under the incongruent condition.
Change scores of the Timed up and go (TUG) test | baseline, posttest (around 12 weeks after baseline)
  The TUG test will be used to assess the mobility and dynamic balance ability. The participants will be required to stand up from a chair, walk 3 meters, turn around, then walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers and frail elderly (Podsiadlo & Richardson, 1991). The test-retest reliability of TUG on individuals with cognitive impairment was excellent.
Change scores of the Dual-task test | baseline, posttest (around 12 weeks after baseline)
  The dual-task tests will be assessed to determine the ability for an individual to perform 2 tasks simultaneously. The investigators will assess the dual-task performance during walking and performing box and block test. The results of the dual-task tests will provide information regarding to whether the 2 tasks compete for the same class of neural resources or one of the tasks can be carried out automatically
Change scores of the Wechsler Adult Intelligence Scale (WAIS) | baseline, posttest (around 12 weeks after baseline)
  Subtests of the Wechsler Adult Intelligence Scale (WAIS) will be used to measure the cognitive functions of an individual. The WAIS have high reliability and validity, and is often used to differentiate individuals with cognitive deficits and those with intact cognitive functions. In addition, WAIS could be used to assess cognitive improvements after an intervention or treatment.
Change scores of the Lawton Instrumental Activities of Daily Living Scale (IADL) | baseline, posttest (around 12 weeks after baseline)
  Assess activities of daily living. There are 8 domains of function measured with the Lawton IADL scale, including ability to use phone,shopping, food preparation, housekeeping, laundering, mode of transportation, responsibility for own medications,and ability to handle finances. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent). For each category, circle the item description that most closely resembles the client's highest functional level (either 0 or 1).
Change scores of the Wechsler Memory Scale (WMS) | baseline, posttest (around 12 weeks after baseline)
  The Wechsler Memory Scale (WMS) was designed to measure different memory functions. The subtests, including Word Lists, and Spatial Span will be used to assess the immediate, delayed, and working memory. Time to administer the WMS subtests is approximately 45 minutes. The total scores range from 0-48 for the immdiate memory, and 0-24 for the delayed memory. Higher values represent a better cognitive functioning.

SECONDARY OUTCOMES:
Change scores of the Community Integration Questionnaire (CIQ) | baseline, posttest (around 12 weeks after baseline)
  The social participation level will be assessed with the Community Integration Questionnaire (CIQ).It contains 15 items to evaluate the degree of integration into each of the three area of family, social network, and productive activities. The total scores range from 0 to 29 with larger numbers indicating better integration.
Change scores of Geriatric Depression Scale (GDS) | baseline, posttest (around 12 weeks after baseline)
  The Geriatric Depression Scale (GDS) - 15 items version is a self-administered questionnaire used to evaluate mood and depressive symptoms. The scores range is 0-15 and a score of 5 or greater taken as a possible indicator of depression.
Change scores of the Everyday Cognition scales (ECog)-12 items | baseline, posttest (around 12 weeks after baseline)
  To detect cognitive and functional decline. The ECog shows promise as a useful tool for the measurement of general and domain-specific everyday functions in the elderly. There are six domains (Everyday Memory, Language, Visuospatial Abilities, Planning, Organization, and Divided Attention) in ECog. Lower scores represent a higher level of function in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Ching yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chuang IC, Chen IC, Wu YR, Li KY. Prediction and mediation analysis for treatment responses to combined cognitive and physical training for older adults. Sci Rep. 2024 May 8;14(1):10571. doi: 10.1038/s41598-024-61407-6. PMID 38720025
- [Derived] Chen IC, Chuang IC, Chang KC, Chang CH, Wu CY. Dual task measures in older adults with and without cognitive impairment: response to simultaneous cognitive-exercise training and minimal clinically important difference estimates. BMC Geriatr. 2023 Oct 16;23(1):663. doi: 10.1186/s12877-023-04390-3. PMID 37845603